CLINICAL TRIAL: NCT02517333
Title: Exploring the Impact and Feasibility of a Pathway to Sport and Long-term Participation in Young People
Acronym: EPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oxford Brookes University (Other)
Collaborators: Sport England (Other); Oxfordshire Sports Partnership (Unknown)
Responsible Party: Principal Investigator, Francesca Liu, Principle Investigator, Oxford Brookes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 140844
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Dyspraxia
Keywords: Motor skill proficiency; movement difficulties; Developmental Coordination Disorder (DCD); Low physical fitness
MeSH Terms: conditions — Apraxias; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proof-of-principle (PoP) (Other): Proof-of-principle phase of the study. All participants undergo the exercise intervention as part of the feasibility.
  1. Screen within Year 9 Class
  2. Targeted recruitment for those scoring in bottom 5th percentile
  3. Invite students to take part in 6-week intervention
  4. Enroll students participating
  5. Pre-intervention assessment
  6. Start 6-week Epic Club gym intervention (1-2 times weekly for 45-60 mins) consisting of 30 min cardiovascular exercise and 25-30 min strength/resistance and weight training
  7. Post-intervention assessment
  8. Exit to longer-term sport/physical activity
  Interventions: Other: EPIC Club

INTERVENTIONS:
Other: EPIC Club — Weekly exercise gym sessions (1-2 times weekly) for 45-60 mins each session. Participants will start with a warm-up of 30 mins cardiovascular training either doing cycling, treadmill running or cross-training. The remainder of the session consists of strength/resistance and weight-training involving leg press, leg extensor, pull downs, kettle bells, dumbbells. Gym sessions aim to involve bursts of high-intensity and monitoring of heart rate (potentially with wrist activity monitors with heart rate monitoring and accelerometers) to identify level of physical activity intensity. Participants will also have the opportunity to engage in 'Have a go' sports days run by the Oxfordshire Sports Partnership.

SUMMARY:
The importance of play and physical activity include its many benefits on positively improving health and well-being, enhancing children's and young people's thinking and performance in school, improving their sleep and enabling confidence and skill building (Janssen and LeBlanc, 2010; Budde et al., 2008; Sallis and Patrick, 1994). However, children with movement difficulties (MD) and physical disabilities are at risk of decreased physical activity and subsequently decreased physical fitness and overall health and well-being as a result. To build upon current findings and to follow-up on a continuing study, looking at the impact (responses) and recovery during and following acute exercise at different intensities in children and adolescents with and without movement difficulties, this next phase aims to provide an intervention to improve fitness levels and health measures and to strategically provide a pathway for longer term participation in physical activity in young people. Implement and evaluate a pathway to sport for 14+ year old young people who do not regularly participate in sport due to Neurodevelopmental conditions, young people presenting with poor coordination and movement, and even children and adolescents with special educational needs. The pathway hopes to promote engagement, participation, inclusion and confidence (EPIC) in sport within local schools and the community through 1) targeted recruitment, 2) confidence and skill building (EPIC Club), 3) connection to sport ('Have a go days') and 4) exit to long term participation.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), physical inactivity is now recognized as the fourth leading risk factor for global mortality for non-communicable diseases, and therefore, supports participation in a variety of physical activities including play, games, sports, planned exercise and resistance training. In accordance, the UK physical activity guidelines for children and young people (ages 5-18) from the Chief Medical Officer (CMO) recommends regular participation in moderate to vigorous physical activity (PA) for at least 60 minutes a day to reduce the risk of children developing cardiovascular conditions later in life. Moreover, the prevalence of neurodevelopmental conditions affecting motor-developmental skills is believed to affect 5-6% of school-aged children and thus, has led to wide interest regarding the physical health and well-being of these children and adolescents due to the lower levels of fitness and participation in PA observed. Participation in PA is often hampered by the limited motor performance capacity of young people with movement difficulties (MD). Furthermore, individuals with poorer motor skills and movement difficulties including Developmental Coordination Disorder (DCD) and cerebral palsy (CP) have reported low energy levels, muscle fatigue and poor physical tolerance as factors contributing to reduced enjoyment, tolerance and participation of PA.

As a consequence, research exploring the fitness and PA patterns of children and adolescents with poor motor proficiency has presented an alarming risk profile for cardiovascular disease, due to higher percentage of body fat, decreased aerobic capacity, and generally decreased participation in PA impacting proper development that may persist into adulthood. Because children with MD are less able to tolerate certain types of exercise and tend to show lower levels of activity, they are at greater risk of developing secondary disorders associated with physical inactivity compared to their typically developing aged peers. Furthermore, although it has been shown that children with MD are willing to push themselves maximally, many fail to exercise hard enough to tax the cardiovascular system, potentially due to and contributing to lower exercise tolerance and lower fitness; all playing a role in a vicious cycle.

Previous work has shown that the condition of a child's muscle strength may be a major contributing factor to exercise (particularly at an intensity high enough to have a training effect). Strength is an essential component of motor skill performance and has become a crucial element incorporated in training interventions. Therefore, developing competence and confidence to perform resistance strength exercise during the developmental years may have important long-term implications for health, fitness and sports performance and even more so for youth with fewer opportunities to do so. In accordance, measures of fitness appear to all be interconnected, with level of motor skill and impairment shown to be related to the maximal oxygen consumption or VO2 peak attained and muscular strength. Exploring the relationships between VO2max and endurance performance in children may provide insights into the basic role of physiologic fitness in dictating physical capacity and for identifying appropriate training regimens in youth. Therefore, it is important to gain a comprehensive picture of the impact of exercise for health and functional measures and to further develop an understanding of the physiological, psychological and social aspects limiting successful long-term PA among children with MD. Implementing interventions that not only involve tasks to improve fitness measures, but also coordination, muscle function and performance, are essential.

Based on a recent Cochrane intervention review looking at school-based PA programs for promoting PA and fitness in children and adolescents aged 6-18 years, the authors suggested that young people exposed to a training intervention spent more time engaged in moderate-to-vigorous PA (with results across studies ranging from 5 - 45 min more a day), spent less time watching television (results ranging from five-60 min less each day) and an improved VO2max (maximal oxygen uptake). However, school-based interventions were not effective in increasing PA rates among adolescents, or in reducing health and fitness markers (i.e. blood pressure, blood cholesterol, BMI and heart rate) (Dobbins et al., 2013), possibly due to insufficient PA intensities. Furthermore, research studying the effects of acute bouts of exercise on cognition has provided compelling evidence for the influence of exercise on working memory. Preliminary results from a current study exploring the impact of acute exercise at high and low exercise intensities is already showing different cognitive responses between individuals with MD compared to their typically developing (TD) peers. Although there is evidence citing the positive impact of increasing PA and play on mood and behaviour, social relationships, sleep, cognition, academic performance and overall well-being, additional research exploring the development, execution, implementation and feasibility of pathways to increase participation and long-term PA and training is warranted. A fitness screening session for a designated year group (i.e. Year 9) will be held at mainstream schools in Oxfordshire. Those scoring in the bottom quintile on fitness tests and/or the motor skill assessment during the screening will be invited to take part in a 6 week training programme (EPIC Club). Participants volunteering to take part will need to attend assessments before and after the training intervention for evaluation of outcome measures including looking at aerobic fitness level, muscles strength, cognitive function and questionnaires focused on self-esteem/self-perception. The aims of EPIC Club are to improve fitness levels, build up confidence and skills and to provide a pathway to sport via 'Have a go' Sports Taster Days held throughout the year. Steering groups and focus groups will also be held inviting the participants, parents and coaches to provide feedback on the progress of the pathway. Moreover, the evaluation of quantitative and qualitative outcome measures needs to be further addressed.

Aims:

1. To deliver a pathway for longer-term participation in physical activity and sport via 1) targeted recruitment, 2) confidence and skill building (EPIC Club), 3) connection to sport ('Have a go days') and 4) exit to long term participation
2. Evaluation and assessment of pathway progress through quantitative and qualitative outcome measures (fitness and physical health measures)
3. To explore impact of pathway program on functioning in other domains, such as cognitive function, performance in school, sleep, self-esteem and social well-being.

Community Benefits:

This study aims to provide a pathway for engagement, participation, inclusion and confidence (EPIC) in sport in young people who do not regularly participate in physical activity and sport due to Neurodevelopmental conditions, young people presenting with poor coordination and movement and/or including individuals with special educational needs. With the rise in obesity and lower physical activity levels, it is important to provide a feasible and meaningful way for young individuals to participate in exercise and sport through community sport activation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to walk with or without support for at least 5 meters, be able to safely take part in two-step instructions.
* GP approval will only be required prior to participation in the training intervention and the assessments if parent/guardian requests so or if the investigators feel there is a need for medical clearance for the child/adolescent to safely participant.
* The participant should be able to mount the cycle ergometer with or without assistance

Exclusion Criteria:

* Any behavioral issues that would prevent safe participation or may put the participant, investigators and others at risk
* Any contraindications to perform maximal exercise
* Individuals suffering from muscular degenerative conditions or with uncontrolled medical conditions (e.g. asthma, diabetes, epilepsy- must be stable and on medication for greater than 12 weeks)

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Fitness Measures | 6 weeks
  Measures are composite and consists of multiple primary outcome measures focused around fitness. Pre- and post-assessments surrounding the EPIC Club gym sessions will seek to monitor changes to fitness measures. The Astrand bike test is a submaximal test of aerobic capacity to predict maximal oxygen uptake based on heart rate and work rate. Arm and leg strength will also be assessed and a motor skill (balance)

SECONDARY OUTCOMES:
Physical activity questionnaire (PAQ-A) and Child Health Utility (9D) Questionnaire | 6 weeks
  Composite of secondary outcome measures for questionnaires including the Physical activity questionnaire (PAQ-A) used to assess physical activity over past 7 days during pre-assessment and the Child Health and Utility (9D) questionnaire focusing on health and overall well-being
  Questionnaire regarding physical activity over the past 7 days
Adherence | 6 weeks
  Number of sessions attended

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, Professor, Principal Investigator — Oxford Brookes University
Locations (5):
- United Kingdom (5):
  - Cherwell School, Oxford
  - CLEAR Unit, Oxford
  - Cheney School, Oxford
  - Wheatley Park School, Oxford
  - The Oxford Academy, Oxford

REFERENCES:
- [Derived] Weedon BD, Liu F, Mahmoud W, Metz R, Beunder K, Delextrat A, Morris MG, Esser P, Collett J, Meaney A, Howells K, Dawes H. The relationship of gross upper and lower limb motor competence to measures of health and fitness in adolescents aged 13-14 years. BMJ Open Sport Exerc Med. 2018 Mar 8;4(1):e000288. doi: 10.1136/bmjsem-2017-000288. eCollection 2018. PMID 29629179